CLINICAL TRIAL: NCT03777865
Title: A PHASE 4, OPEN-LABEL, SINGLE-ARM, MULTICENTER STUDY TO DESCRIBE THE SAFETY OF 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN CHILDREN 6 TO 17 YEARS OF AGE IN INDIA
Brief Title: Study To Describe The Safety Of 13-valent Pneumococcal Conjugate Vaccine In Children 6 To 17 Years Of Age In India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1851190; 13VPNC 6 TO 17 YEARS IN INDIA (Other: Alias Study Number); 2019-000890-21 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2018-12-17 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 13vPnC provided as a 0.5-mL dose in a prefilled syringe (Experimental): All subjects receive a single dose (0.5mL) of 13vPnC
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 13vPnC — All subjects receive a single dose (0.5mL) of 13vPnC

SUMMARY:
This is a Phase 4, open-label, single-arm, multicenter study in which subjects 6 to 17 years of age will receive 1 dose of 13vPnC.

DETAILED DESCRIPTION:
A Phase 4, open-label, single-arm, multicenter study to describe the safety of 13-valent Pneumococcal Conjugate Vaccine in children 6 to 17 years of age in India.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject's parent(s)/legal guardian(s) has/have been informed of all pertinent aspects of the study.

   Note: The subject's assent may also be required depending on local requirements.
2. Healthy male or female children 6 to 17 years of age at the time of vaccination.
3. Parent(s)/legal guardian(s)/child willing and able to comply with scheduled visits, treatment plan, and other study procedures.
4. Male subject not able to father children, male subject who is able to father children and willing to use a highly effective method of contraception, female subject not of childbearing potential, or female subject of childbearing potential and at risk for pregnancy who is willing to use a highly effective method of contraception.

Note: Female subjects of childbearing potential are defined as female subjects 9 years old or have experienced menarche, whichever is earlier, and who are anatomically and functionally able to conceive.

Exclusion Criteria:

1. Child who is a family member of:

   * Investigator site staff members directly involved in the conduct of the study;
   * Site staff members otherwise supervised by the investigator;
   * Pfizer employees directly involved in the conduct of the study.
2. Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation. Participation in observational studies is permitted.
3. History of severe adverse reaction, including hypersensitivity such as anaphylaxis, associated with a vaccine or vaccine component.
4. Contraindication to vaccination with pneumococcal conjugate vaccines (refer to local package insert).
5. Previous vaccination with licensed or investigational pneumococcal vaccine.
6. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
7. History of culture-proven invasive disease caused by S pneumoniae.
8. Major known congenital malformation or serious chronic disorder.
9. Known or suspected immune deficiency or suppression.
10. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
11. Pregnant females; breastfeeding females; fertile males and females of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- India (4):
  - Manipal Hospital / Department of Pediatrics, Bengaluru, Karnataka
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Christian Medical College, Ludhiana, Punjab
  - Kanchi Kamakoti CHILDS Trust Hospital, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851190

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 1 country from 14 December 2018 to 17 April 2019. A total of 100 participants were enrolled.
Groups:
- 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine: Participants received a single dose of 0.5 milliliter (mL) 13vPnC vaccine, intramuscularly on Day 1.
Period: Overall Study
Arm/Group | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received 1 dose of an investigational product.
Groups:
- 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine: Participants received a single dose of 0.5 mL 13vPnC vaccine, intramuscularly on Day 1.
Arm/Group | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.28 (2.985)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 100
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Local Reactions by Severity Within 7 Days After Vaccination
Description: Local reactions (redness, swelling and pain [tenderness]) at the 13vPnC injection site were monitored daily for 7 days after vaccination. Redness and swelling were measured and recorded in a measuring device units. 1 measuring device unit=0.5 centimeter (cm). Redness and swelling were graded as; any (any redness or swelling at the injection site), mild (1 to 4 measuring device units = 0.5 to 2.0 cm), moderate (5 to 14 measuring device units = 2.5 to 7.0 cm) and severe (greater than [>]14 measuring device units = >7.0 cm). Pain (tenderness) at injection site was categorized as; any: any pain at the injection site, mild: did not interfere with activity, moderate: interfered with activity and severe: prevented daily activity.
Time Frame: Within 7 days after vaccination on Day 1 (up to Day 7)
Population: The safety population included all participants who received 1 dose of an investigational product. Here, "Overall Number of Participants Analyzed"=Participants evaluable for this outcome measure and "Number Analyzed"=Participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine
Number analyzed (Participants) | 92
percentage of participants
  Redness: Any: number analyzed (Participants) | 74
  Redness: Any | 14.9 [7.7 to 25.0]
  Redness: Mild: number analyzed (Participants) | 74
  Redness: Mild | 14.9 [7.7 to 25.0]
  Redness: Moderate: number analyzed (Participants) | 74
  Redness: Moderate | 0 [0.0 to 4.9]
  Redness: Severe: number analyzed (Participants) | 74
  Redness: Severe | 0 [0.0 to 4.9]
  Swelling: Any: number analyzed (Participants) | 74
  Swelling: Any | 17.6 [9.7 to 28.2]
  Swelling: Mild: number analyzed (Participants) | 74
  Swelling: Mild | 17.6 [9.7 to 28.2]
  Swelling: Moderate: number analyzed (Participants) | 74
  Swelling: Moderate | 0 [0.0 to 4.9]
  Swelling: Severe: number analyzed (Participants) | 74
  Swelling: Severe | 0 [0.0 to 4.9]
  Pain: Any: number analyzed (Participants) | 91
  Pain: Any | 67.0 [56.4 to 76.5]
  Pain: Mild: number analyzed (Participants) | 91
  Pain: Mild | 45.1 [34.6 to 55.8]
  Pain: Moderate: number analyzed (Participants) | 91
  Pain: Moderate | 19.8 [12.2 to 29.4]
  Pain: Severe: number analyzed (Participants) | 91
  Pain: Severe | 2.2 [0.3 to 7.7]

2. Primary Outcome: Percentage of Participants Reporting Systemic Events by Severity Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue(tiredness), headache, muscle pain, joint pain, vomiting and diarrhea. Fever: greater than or equal to (>=) 38.0 degrees Celsius (C), >=38.0 degrees C to <=38.4 degrees C, >=38.5 to <=38.9 degrees C, 39.0 to 40.0 degrees C, > 40.0 degrees C. Fatigue, headache, muscle pain and joint pain graded as any (any fatigue, headache, muscle pain, joint pain), mild(did not interfere with activity), moderate(some interference with activity) or severe(prevented daily routine activity). Vomiting was graded as any (any vomiting), mild (1-2 times in 24 hours [hrs.]), moderate(>2 times in 24 hrs.) or severe (required intravenous hydration). Diarrhea was graded as any(any diarrhea), mild (2-3 loose stools in 24 hrs.), moderate(4-5 loose stools in 24 hrs.) or severe(>=6 loose stools in 24 hrs.)
Time Frame: Within 7 days after vaccination on Day 1 (up to Day 7)
Population: The safety population included all participants who received 1 dose of an investigational product. Here "Overall Number of Participants Analyzed"=Participants evaluable for this outcome measure and "Number Analyzed"=Participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine
Number analyzed (Participants) | 83
percentage of participants
  Fever: >=38 degrees C: number analyzed (Participants) | 73
  Fever: >=38 degrees C | 4.1 [0.9 to 11.5]
  Fever: >=38 degrees C to <=38.4 degrees C: number analyzed (Participants) | 73
  Fever: >=38 degrees C to <=38.4 degrees C | 1.4 [0.0 to 7.4]
  Fever:>=38.5 degrees C to <=38.9 degrees C: number analyzed (Participants) | 73
  Fever:>=38.5 degrees C to <=38.9 degrees C | 2.7 [0.3 to 9.5]
  Fever:>=39.0 degrees C to <=40.0 degrees C: number analyzed (Participants) | 73
  Fever:>=39.0 degrees C to <=40.0 degrees C | 0 [0.0 to 4.9]
  Fever: >40.0 degrees C: number analyzed (Participants) | 73
  Fever: >40.0 degrees C | 0 [0.0 to 4.9]
  Fatigue: Any: number analyzed (Participants) | 77
  Fatigue: Any | 31.2 [21.1 to 42.7]
  Fatigue: Mild: number analyzed (Participants) | 77
  Fatigue: Mild | 22.1 [13.4 to 33.0]
  Fatigue: Moderate: number analyzed (Participants) | 77
  Fatigue: Moderate | 6.5 [2.1 to 14.5]
  Fatigue: Severe: number analyzed (Participants) | 77
  Fatigue: Severe | 2.6 [0.3 to 9.1]
  Headache: Any: number analyzed (Participants) | 76
  Headache: Any | 25.0 [15.8 to 36.3]
  Headache: Mild: number analyzed (Participants) | 76
  Headache: Mild | 15.8 [8.4 to 26.0]
  Headache: Moderate: number analyzed (Participants) | 76
  Headache: Moderate | 6.6 [2.2 to 14.7]
  Headache: Severe: number analyzed (Participants) | 76
  Headache: Severe | 2.6 [0.3 to 9.2]
  Muscle pain: Any: number analyzed (Participants) | 77
  Muscle pain: Any | 27.3 [17.7 to 38.6]
  Muscle pain: Mild: number analyzed (Participants) | 77
  Muscle pain: Mild | 20.8 [12.4 to 31.5]
  Muscle pain: Moderate: number analyzed (Participants) | 77
  Muscle pain: Moderate | 3.9 [0.8 to 11.0]
  Muscle pain: Severe: number analyzed (Participants) | 77
  Muscle pain: Severe | 2.6 [0.3 to 9.1]
  Joint pain: Any: number analyzed (Participants) | 77
  Joint pain: Any | 13.0 [6.4 to 22.6]
  Joint pain: Mild: number analyzed (Participants) | 77
  Joint pain: Mild | 3.9 [0.8 to 11.0]
  Joint pain: Moderate: number analyzed (Participants) | 77
  Joint pain: Moderate | 7.8 [2.9 to 16.2]
  Joint pain: Severe: number analyzed (Participants) | 77
  Joint pain: Severe | 1.3 [0.0 to 7.0]
  Vomiting: Any: number analyzed (Participants) | 73
  Vomiting: Any | 9.6 [3.9 to 18.8]
  Vomiting: Mild: number analyzed (Participants) | 73
  Vomiting: Mild | 8.2 [3.1 to 17.0]
  Vomiting: Moderate: number analyzed (Participants) | 73
  Vomiting: Moderate | 1.4 [0.0 to 7.4]
  Vomiting: Severe: number analyzed (Participants) | 73
  Vomiting: Severe | 0 [0.0 to 4.9]
  Diarrhea: Any: number analyzed (Participants) | 73
  Diarrhea: Any | 4.1 [0.9 to 11.5]
  Diarrhea: Mild: number analyzed (Participants) | 73
  Diarrhea: Mild | 2.7 [0.3 to 9.5]
  Diarrhea: Moderate: number analyzed (Participants) | 73
  Diarrhea: Moderate | 1.4 [0.0 to 7.4]
  Diarrhea: Severe: number analyzed (Participants) | 73
  Diarrhea: Severe | 0 [0.0 to 4.9]

3. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event. Treatment-emergent were events between first dose of study drug and up to 1 month that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: up to 1 month after vaccination on Day 1
Population: The safety population included all participants who received 1 dose of an investigational product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine
Number analyzed (Participants) | 100
percentage of participants
  AEs | 75.0 [65.3 to 83.1]
  SAEs | 1.0 [0.0 to 5.4]

ADVERSE EVENTS:
Time Frame: up to 1 month after vaccination on Day 1
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study.
Arm/Group | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 75/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine (N=100)
Hepatitis acute (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13-Valent Pneumococcal Conjugate (13vPnC) Vaccine (N=100)
Diarrhoea (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (General disorders) | 3/73 — Number of participants exposed = number of participants evaluable for the adverse event.
Vomiting (General disorders) | 7/73 — Number of participants exposed = number of participants evaluable for the adverse event.
Fatigue (General disorders) | 24/77 — Number of participants exposed = number of participants evaluable for the adverse event.
Fever (General disorders) | 3/73 — Number of participants exposed = number of participants evaluable for the adverse event.
Joint pain (General disorders) | 10/77 — Number of participants exposed = number of participants evaluable for the adverse event.
Muscle pain (General disorders) | 21/77 — Number of participants exposed = number of participants evaluable for the adverse event.
Pain at the injection site (Skin and subcutaneous tissue disorders) | 61/91 — Number of participants exposed = number of participants evaluable for the adverse event.
Redness (Skin and subcutaneous tissue disorders) | 11/74 — Number of participants exposed = number of participants evaluable for the adverse event.
Swelling (Skin and subcutaneous tissue disorders) | 13/74 — Number of participants exposed = number of participants evaluable for the adverse event.
Headache (General disorders) | 19/76 — Number of participants exposed = number of participants evaluable for the adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03777865/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03777865/SAP_001.pdf